CLINICAL TRIAL: NCT06607705
Title: Fluctuations of the Intraocular Pressure in Surgically Treated Glaucoma Patients with IStent Inject W by a Contact Lens Sensor
Brief Title: Changes in Eye Pressure in Glaucoma Patients Treated with Istent Inject W, Monitored by a Contact Lens Sensor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Privada Mon Clinic Barcelona (Other)
Collaborators: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GLAUKOS
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma Eye
Keywords: intraocular pressure (IOP); glaucoma; cataract; ophthalmology; Contact Lens Sensor (CLS); Glaucoma surgery; iStent inject W; Sensimed Triggerfish
MeSH Terms: conditions — Glaucoma; Cataract

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-randomized, controlled, single country pre-post intervention study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery required glaucoma (Experimental): Treatment group
  Interventions: Device: Monitoring with contact lens sensor
- Medically controlled glaucoma (Experimental): Control group
  Interventions: Device: Monitoring with contact lens sensor

INTERVENTIONS:
Device: Monitoring with contact lens sensor — Monitoring with contact lens sensor at 1-month pre-intervention visit
Device: Monitoring with contact lens sensor — Monitoring with contact lens sensor at 1-month post-intervention visit
  Arms: Surgery required glaucoma
Device: Monitoring with contact lens sensor — Monitoring with contact lens sensor at 3-months post-intervention visit

SUMMARY:
The purpose of this study is to compare the IOP-related fluctuations using the CLS (contact lens sensor) Sensimed Triggerfish in glaucoma patients before and after glaucoma surgery with iStent inject W under physiological conditions and compare these results with a control group of glaucoma patients treated only with hypotensive medical treatment requiring cataract surgery.

DETAILED DESCRIPTION:
This is a prospective controlled pre-post intervention study conducted at a Hospital Clínic of Barcelona, a university hospital in Barcelona, Spain. This study will be adhered to the tenets of the Declaration of Helsinki. Informed patient consent and approval by the Institutional Review Board will be obtained prior to study commencement. Study duration is expected to be around 12 months, recruitment period would last between 6 to 8 months and study is expected to be finalized by Jun 2025.

The study will recruit consenting adults (over 18 years old) with unilateral or bilateral primary open-angle glaucoma (POAG) without previous eye surgery, treated with topical anti-glaucoma medications, who need glaucoma surgery with iStent inject W. The investigators will include patients with isolate iStent surgery and patients with combined cataract and iStent surgery. In cases of bilateral glaucoma, the two eyes of the same patient may be included consecutively.

One month prior to glaucoma surgery with iStent inject W, subjects will wear the CLS for 24 hours without changing the regimen of anti-glaucoma eye drops. The CLS will be placed on the subject's eye by an ophthalmologist in the clinic after a slit lamp examination and keratometry to determine the corneal curvature for selection of the appropriate CLS base curve. The subjects will then return home and carry on their routine activities (both indoor and outdoor), apart from showering or swimming (as the device cannot be in contact with water). Subjects will continue the same regimen of anti-glaucoma eye drops and slept in their habitual position at night. Each subject will carry a logbook to record sleeping and medication instillation times during the 24-hour period. After 24 hours, the subject will return to the clinic to have the contact lens removed followed by a slit lamp examination. The data recorded by the CLS will be uploaded into a computer database. Goldmann applanation tonometry (GAT) will be perform before and after each CLS wear by a single observer. At 1-month (n=9/44) and 3-month (n=44) post-glaucoma surgery with iStent implant, patients will wear the CLS in the same eye that received the first CLS recording. As before, the CLS will be removed 24 hours later. To extend the follow-up to 3 months after surgery will allow us to corroborate that the effects of the surgery on fluctuations of IOP for 24 hours are maintained over time. In the control group (n=10) , a first monitoring with CLS will be carried out one month before cataract surgery, and a second monitoring will be carried out 3 months after this cataract surgery, without us having introduced any changes in their hypotensive medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients (over 18 years old) with an initial diagnosis of POAG requiring an indication from the patient chart of an untreated IOP of over 21 mm Hg. Diagnosis of NTG requiring an untreated mean diurnal IOP of over 21 mm Hg from diagnosis to enrollment, indicated by the patient chart. Ocular hypertension is defined as a condition in which the IOP was greater than 21 mm Hg in the absence of glaucomatous defects in visual field testing, the normal appearance of the optic disc and nerve fiber layer, anatomic normality, open angles in gonioscopy, and the absence of ocular conditions contributing to the elevation of pressure, such as narrow angles, neovascular conditions, and uveitis.
* Adult Patients (over 18 years old ) diagnosed with POAG and NTG are defined as those with open normal appearing angles, typical glaucomatous optic atrophy (i.e., neural rim thinning, notching, saucerization, or nerve fiber layer disc haemorrhage), and typical glaucomatous visual field damage (i.e., arcuate, paracentral scotoma, or nasal step).
* Adult Patients (age over 18 years old ):

with unilateral or bilateral open-angle glaucoma (POAG) without previous eye surgery, treated with topical anti-glaucoma medications, who need glaucoma surgery with iStent inject W. The investigators will include patients with isolate iStent surgery and patients with combined cataract and iStent surgery. In cases of bilateral glaucoma, the two eyes of the same patient may be included consecutively.

For the control group only: Patients with topical hypotensive glaucoma treatment requiring cataract surgery.

Exclusion Criteria:

* Age under 18 years
* Visual defects attributable to nonglaucomatous conditions, primary angle closure glaucoma, neovascular glaucoma, history of ocular trauma, retinal disease or ocular inflammation, and laser therapy or secondary glaucoma.
* The patients have to meet best-corrected Snellen visual acuity of under 0.3 and spherical equivalent of under 6 diopter.
* We will not include patients with previous ocular surgery, except cataract surgery performed at least 6 months prior to the inclusion date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
IOP-related fluctuation over a 24- hour period | 24 hours during 1-month pre-intervention visit, 24 hours during 1-month post-intervention visit and 24 hours during 3-month post-intervention visit
  The amplitude of the cosine curve is a parameter based on the cosine model fitted to the CLS data. The amplitude is the difference between the maximum and minimum values of the cosine-fit curve divided by 2. This is an overall estimate of the magnitude of signal oscillation during the tested period. The cosinor model represents the actual amplitude of IOP-related fluctuation over a 24- hour period and is most representative of IOP-related changes.
  IOP-related fluctuations will be calculated based on the GAT IOP measured at baseline and at each visit during the study.
  Control group will not be monitored in the 1-month visit.
CLS increase and decrease rates | 24 hours during 1-month pre-intervention visit, 24 hours during 1-month post-intervention visit and 24 hours during 3-month post-intervention visit
  CLS (Contact Lens Sensor) increase and decrease rates (change in CLS units/ change in time): maximum
  Control group will not be monitored in the 1-month visit.
CLS increase and decrease rates | 24 hours during 1-month pre-intervention visit, 24 hours during 1-month post-intervention visit and 24 hours during 3-month post-intervention visit
  CLS (Contact Lens Sensor) increase and decrease rates (change in CLS units/ change in time): minimum.
  Control group will not be monitored in the 1-month visit.
CLS increase and decrease rates | 24 hours during 1-month pre-intervention visit, 24 hours during 1-month post-intervention visit and 24 hours during 3-month post-intervention visit
  CLS (Contact Lens Sensor) increase and decrease rates (change in CLS units/ change in time): median.
  Control group will not be monitored in the 1-month visit.
CLS increase and decrease rates | 24 hours during 1-month pre-intervention visit, 24 hours during 1-month post-intervention visit and 24 hours during 3-month post-intervention visit
  CLS (Contact Lens Sensor) increase and decrease rates (change in CLS units/ change in time): mean.
  Control group will not be monitored in the 1-month visit.
Sleep-to-wake slope | 24 hours during 1-month pre-intervention visit, 24 hours during 1-month post-intervention visit and 24 hours during 3-month post-intervention visit
  Calculation of sleep-to-wake slope.
  Control group will not be monitored in the 1-month visit.
Wake-to-sleep slope | 24 hours during 1-month pre-intervention visit, 24 hours during 1-month post-intervention visit and 24 hours during 3-month post-intervention visit
  Calculation of wake-to-sleep slope.
  Control group will not be monitored in the 1-month visit.
Number of peaks of IOP-related fluctuations | 24 hours during 1-month pre-intervention visit, 24 hours during 1-month post-intervention visit and 24 hours during 3-month post-intervention visit
  Number of peaks: over 24 hours, inferior to 30 minutes, superior to 90mVeq.
  Control group will not be monitored in the 1-month visit.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Institut Català de Retina, Barcelona, Spain
  - Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No